CLINICAL TRIAL: NCT05388864
Title: A Multi-Component Intervention to Strengthen Families With Adverse Childhood Experiences (ACEs)
Brief Title: Building Resilient Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5180358
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Adverse Childhood Experiences
Keywords: adverse childhood experiences; pediatrics; prevention; preventive health services; quality improvement; childhood abuse and neglect

STUDY DESIGN:
Intervention Model Description: Pediatric providers are randomized to training on the intervention or usual well-child care. Three groups of patients are recruited to evaluate the efficacy of the intervention: 1) Usual well-child care for children with no ACEs; 2) Usual well-child care for children with ACEs; and 3) Well-child care by providers trained in the intervention.
Who Masked: Participant
Masking Description: The pediatric patients, their caregivers and teachers are blinded to arm type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Three-Tier Model (Experimental): 130 children with ACEs who received well-child care by a trained provider will be enrolled in this group.
  Interventions: Behavioral: Three-Tier Model
- Comparison Group (No Intervention): 80 children without ACEs who received usual well-child care will be enrolled in this group.
- Control Group (No Intervention): 130 children with ACEs who received usual well-child care will be enrolled in this group.

INTERVENTIONS:
Behavioral: Three-Tier Model — Families in the intervention will be counseled by a pediatric provider about ACEs, resilience, stress management, and healthy relationships. Families will also be referred to community health workers and parenting educators.
  Arms: Three-Tier Model

SUMMARY:
Prior research suggests that it is possible to improve health outcomes in children with ACEs through multi-component interventions. The challenge for most communities is that health and education systems are fragmented and fail to accommodate families based upon different levels of need. This study utilizes cross-sectoral partnerships to mobilize three vectors (pediatricians, community health workers and parenting educators) to optimize the delivery of vital information and resources to a diverse population of families with ACEs. All vectors are trained in an evidence-informed curriculum to strengthen families and build youth resilience. The study design is a randomized controlled trial of 340 families of children between the ages of 3 to 11 who are generally healthy and have recently seen a pediatrician for a well-child visit.

To evaluate the efficacy of this intervention, pediatric patients are invited to participate in repeat evaluations within 2 weeks, 3 months, 6 months, and 12 months after their well-child visit. The study will evaluate the following: 1) the association between Child-ACE scores and biomarkers of toxic stress at baseline in children age 3-11 years old; 2) whether the intervention reduces toxic stress and child health and psychosocial problems at follow-up for children with ACEs compared to usual well-child care for children with ACEs; and 3) the impact of mediating and moderating variables. These results will demonstrate that for families with ACEs the intervention will decrease toxic stress associated with ACEs, improve health outcomes, and reduce health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-11
* Seen for a well-child visit at a participating pediatric clinic

Exclusion Criteria:

* < 3 years or >11 years of age
* Significant congenital medical problems
* Previous participation in parenting program (last 12 months)
* Sibling enrollment in current study

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Child Allostatic Load Index | Change between baseline and visit 4 (1-year post-enrollment)
  A composite measurement that combines biometric data, neuroendocrine and immune markers, and executive function to determine whether the intervention lowers physiologic stress for children with ACEs. Each group will be followed over one year and growth curves will be analyzed to compare change in physiologic stress between baseline and final follow-up.

SECONDARY OUTCOMES:
Pediatric Symptom Checklist (PSC) | Change between baseline and visit 4 (1-year post-enrollment)
  The Pediatric Symptom Checklist is a psychosocial screen designed to indicate psychological impairment.
  For participants ages 3-5, a total score of 24 indicates psychological impairment.
  For participants ages 6-11, a total score of 28 indicates psychological impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Marie-Mitchell, MD, PhD, MPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No